CLINICAL TRIAL: NCT01282567
Title: Preliminary Study for the Artificial Pancreas Project : Determination of a Tuning Strategy of Metabolic Profiles
Brief Title: Study for the Artificial Pancreas Project : Determination of a Tuning Strategy of Metabolic Profiles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2010-A01455-34; LOC/10-18
Record Dates: First submitted 2011-01-20; First posted 2011-01-25 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Specimen Collection

ARMS (1):
- diabetic patients (Other)
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — The study will be proposed to four patients hospitalized in the Diabetes Unit for a glucidic fast test carried out during 24 hours (lunch, dinner and breakfast). Blood samples will be taken every 20 minutes during 6 hours and 40 minutes to measure plasma insulin concentration and blood glucose. T0 will correspond to the first modification of the insulin basal flow (in more or less) or to the first insulin bolus corrector, usually administered if capillary blood glucose reaches 1.8 g/l. The capillary blood glucose monitoring will be performed every two hours by the nurse.

SUMMARY:
The Artificial Pancreas Project developed by SUPELEC and the University Hospital of Rennes is focused on the evaluation of an original control algorithm that computes appropriate subcutaneous insulin infusion in response to continuous glucose measurements The results during a 24-hour closed-loop period will be compared with those of the open-loop. The implementation of this algorithm named Error Dynamics Shaping (EDS) requires as a preliminary a phase of identification of the parameters of the model (insulin pharmacokinetics and effect on glucose metabolism) followed by a phase of optimization i.e. a personalized adjustment of the damping parameters of EDS.

The present study aims to formalize this procedure of identification/optimization of the parameters of the model and controller EDS. They will be determined in type -1 diabetic patients using insulin therapy and under conditions free from disturbances such as those generated by the glucidic meals, i.e. during a period of glucidic fast. Three variables will determine this procedure: blood glucose, insulin concentration and insulin doses.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetic patients (age : 18-70)
* Diabetes duration higher than three years
* Insulin pump with Humalog®
* Hospitalized for a 24-hour glucidic fast test
* Written informed consent

Exclusion Criteria:

* Pregnancy or nursing
* Acute infectious disease
* Corticoid treatment
* Creatinine clearance <40 ml/mn
* Patients using Apidra® or Novorapid®
* People major being the object of a legal protection (safeguard of justice, supervision, trusteeship)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Dosage of plasma insulin concentration and blood glucose every 20 minutes during 6 hours and 40 minutes | 3 months
  Identification of the eight parameters of the model including the five parameters of the glucose/insulin metabolism (p1, p2, p3, GB and Ib) and the three parameters of the model of subcutaneous insulin absorption Optimization of the four damping parameters of EDS. These coefficients can be tuned to adjust the damping degree of the error dynamics.
  These procedures of identification and optimization will be carried out under Matlab® and Simulink®.

CONTACTS AND LOCATIONS:
Overall Officials: jean-yves poirier, Principal Investigator — Rennes University Hospital; isabelle guilhem, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France